CLINICAL TRIAL: NCT04572009
Title: Validation of a Biomathematical Model to Help Identify the Parameters of Flexible Insulin Therapy: Monocentric, Controlled, Randomized and Prospective Pilot Clinical Study in Patients With Type 1 Diabetes.
Brief Title: Validation of a Biomathematical Model to Help Identify the Parameters of Flexible Insulin Therapy
Acronym: ModIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC20_0278
Record Dates: First submitted 2020-09-22; First posted 2020-10-01 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes mellitus; biomathematical model; Flexible insulin therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented physician (Experimental): Medical decision assisted by the bio-mathematical model to define the parameters of flexible insulin therapy based on data from a continuous glucose measurement record.
  Interventions: Other: Bio-mathematical model
- Control (Placebo Comparator): Unassisted medical decision to define the parameters of flexible insulin therapy based on data from a continuous glucose measurement record.
  Interventions: Other: Without bio-mathematical model

INTERVENTIONS:
Other: Bio-mathematical model — bio-mathematical model to help the physician identify the parameters of flexible insulin therapy (basal rate, insulin sensitivity, carbohydrate ratios)
  Arms: Augmented physician
Other: Without bio-mathematical model — No bio-mathematical model to help the physician identify the parameters of flexible insulin therapy (basal rate, insulin sensitivity, carbohydrate ratios)
  Arms: Control

SUMMARY:
Type 1 diabetes is an autoimmune disease that requires daily treatment with insulin. The use of subcutaneous pumps for continuous insulin delivery has been an important advance for diabetic patients. The evolution of technologies through the miniaturization of insulin pumps and the advent of continuous glucose sensors has made it possible to understand the development of the artificial pancreas. Several teams are working on the development of an artificial pancreas with considerable progress in closed-loop insulin delivery, particularly during the night.

The Laboratory of Digital Sciences of Nantes has developed a new bio-mathematical model describing the glucose-insulin dynamics, closer to the physiological reality of patients with type 1 diabetes. This model allows firstly to identify the parameters of flexible insulin therapy (basal rate, insulin sensitivity, carbohydrate ratios).

The objective of this study is to test the relevance of this bio-mathematical model to help the physician identify the parameters of flexible insulin therapy (basal rate, insulin sensitivity, carbohydrate ratios).

DETAILED DESCRIPTION:
This is an open randomized pilot clinical study, comparing the effectiveness of medical decision assisted by this bio-mathematical model ("augmented physician") versus unassisted medical decision, to define the parameters of flexible insulin therapy based on data from a continuous glucose measurement record for 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with type 1 diabetes for at least two years with an indication for sensor placement,
2. Patient patient with at least 6 months of external insulin pump therapy and using the Medtronic 640G pump with or without the Enlite® System.
3. Patient having at least 6 months experience of flexible insulin therapy,
4. Patient with HbA1c <10% (less than 4 months' duration of testing in a medical laboratory or equivalent),
5. Patient who has been wearing a Continuous Glucose Monitoring device for at least 3 months,
6. Adult patient,
7. Patient affiliated to a Social Security or equivalent,
8. Patient who has signed Informed Consent Form.

Exclusion Criteria:

1. Patient with type 2 diabetes or secondary diabetes
2. Patient with any serious medical condition that may affect participation in the study,
3. Patient benefiting from a legal protection measure,
4. Woman who is pregnant or likely to become pregnant during the course of the study, i.e., a lack of effective contraception in women of childbearing age,
5. Breastfeeding,
6. Psychological and/or physical condition that may affect the proper monitoring of study procedures,
7. Severe hypoglycemia leading to convulsions or loss of consciousness within the last 12 months,
8. Decreased hypoglycemic feelings (as judged by the clinician),
9. Impaired renal function (creatinine clearance calculated by CKD-EPI < 30mL/min),
10. Patient who has had a pancreas transplant or pancreatic islets,
11. Persons with severe uncorrected hearing and/or visual acuity problems,
12. Insulin resistance defined by daily insulin requirements > 1 U/kg/day in the week prior to inclusion,
13. Patient treated with oral corticosteroid therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-10-04 (Actual)

PRIMARY OUTCOMES:
percentage of time in glycemic target | 4 weeks
  percentage of time in glycemic target (70-180 mg/dL) during the four weeks following medical consultation where the parameters of flexible insulin therapy are estimated by the physician, either conventionally or with the help of the bio-mathematical model, and parameterized in the insulin pump.

SECONDARY OUTCOMES:
Coefficient of variation of glucose | 75 days
  Hypoglycemic readings < 0.7 g/L, Time below 0.7 g/L, Time above 1.8 g/L
Frequency of severe hypoglycemia | 75 days
  Frequency of severe hypoglycemia (requiring the intervention of a third party)
Robustness of the model | 75 days
  for each glycemic holter, identification of the model from the first 3 days of recording and comparison during the last 3 days of the predicted results with the observed glucose levels. And comparison, in the "delayed modelling" arm, of the doses estimated by the diabetologist and the doses estimated from the model.
assessment of patient compliance | 75 days
  evaluation of the difference between the theoretical doses recommended following modelling and the actual doses given by the patient
assessment of patient acceptance | 75 days
  Quality of life questionnaire SF36
the average time of medical consultation in each group. | 75 days
  Duration of the consultation
changes in heart rate over time | 75 days
changes in activity over time | 75 days

CONTACTS AND LOCATIONS:
Overall Officials: Lucy CHAILLOUS, Dr, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France

REFERENCES:
- [Derived] Scharbarg E, Greck J, Le Carpentier E, Chaillous L, Moog CH. A metamodel-based flexible insulin therapy for type 1 diabetes patients subjected to aerobic physical activity. Sci Rep. 2022 May 16;12(1):8017. doi: 10.1038/s41598-022-11772-x. PMID 35577814